CLINICAL TRIAL: NCT03082027
Title: Pre-operative Sonographic Assessment of The Median Nerve in Carpal Tunnel Syndrome. Does it Affect The Operative Procedure?
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Allam, Lecturer of orthopaedic surgery, Minia University
Other Study IDs: Minia university
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: CTS
Keywords: ultrasonography; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ultrasonography: diagnostic tool
  Interventions: Diagnostic Test: ultrasonography
- operative release
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — ultrasonography of median nerve

SUMMARY:
Sonographic Assessment of The Median Nerve in Carpal Tunnel Syndrome to assess the surgical importance and added value of superficial ultrasonography in assessment of the median nerve in CTS.

DETAILED DESCRIPTION:
Abstract Objective: To assess the surgical importance and added value of superficial ultrasonography in assessment of the median nerve in CTS.

Methods: The study was conducted on thirty patients with CTS with electrophysiological confirmation; twelve males and eighteen females with mean age 43.93±4.51 (range 35-52y), and another thirty normal subjects; fifteen males and fifteen females, with their mean age 36.7±4.86 (range 29-45y). The cross sectional area (CSA) and flattening ratio (FR) at different levels were measured on both groups. Data from the study and control groups were compared. The accuracy of the ultrasonographic diagnostic criteria for CTS was evaluated using receiver operating characteristic (ROC) analysis. All the patients had surgical carpal tunnel release and the operative details were correlated with the ultrasonographic data.

ELIGIBILITY:
Inclusion Criteria:

* Carpal tunnel syndrome

Exclusion Criteria:

* bifid median nerve, carpal tunnel mass lesions, persistent median artery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Thirty patients diagnosed as CTS were referred from the orthopedic clinics Another thirty healthy asymptomatic persons were included in this study as a control group
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
cross sectional area | three minutes
flattening ratio | three minutes

SECONDARY OUTCOMES:
cross sectional area difference | three minutes

IPD SHARING:
Plan to Share IPD: Undecided